CLINICAL TRIAL: NCT05090475
Title: Evaluating Hospital Educator-led Academic Detailing on Improving Antibiotic Prescribing in Primary Healthcare: a Feasibility Study
Brief Title: Implementation of Academic Detailing Interventions on Prescribing of Antimicrobial Drugs in Primary Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital Koprivnica (Other)
Collaborators: Koprivnica Križevci County (Unknown); Interdisciplinary section for the control of antibiotic resistance (ISKRA) (Unknown)
Responsible Party: Principal Investigator, Darija Kuruc Poje, Head of hospital pharmacy, Clinical pharmacist, General Hospital Koprivnica
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: hospital A-team_primary care
Record Dates: First submitted 2021-07-06; First posted 2021-10-22 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Upper Respiratory Tract Infections; Acute Respiratory Tract Infection; Viral Infection
Keywords: Antimicrobial resistance; Hospital A-team; Academic detailing intervention; Antimicrobial prescribing; Primary care
MeSH Terms: conditions — Respiratory Tract Infections; Virus Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group in Koprivnica Križevci County (Experimental): Hospital A-team provided academic detailing intervention to primary care physicians in Koprivnica Križevci county who agree to participate
  Interventions: Behavioral: Academic detailing intervention
- Control group in Koprivnica Križevci county (No Intervention): Primary care physicians in Koprivnica Križevci county who did not agree to participate in academic detailing intervention
- Control group in Bjelovar Bilogora county (No Intervention): Primary care physicians in Bjelovar Bilogora county without the academic detailing intervention

INTERVENTIONS:
Behavioral: Academic detailing intervention — Academic detailing or educational outreach is a method based on scientific data with the help of educated A-team members in the form of direct (face-to-face) interactions, prescribing practices change and adherence improves according to the application of currently valid therapeutic guidelines
  Arms: Experimental group in Koprivnica Križevci County

SUMMARY:
World increase in mortality from consequences of antimicrobial resistance (AMR) represents a significant public health problem. Irrational prescribing of antimicrobial drugs (AMD) in general population is one of the main causes of development AMR. This is also contributed by fact that up to 90% of total antimicrobial consumption in Europe is related to the general population. Problem of AMR has been recognized by World Health Organization and Council of European Union, which support the establishment of the antimicrobial stewardship team (A-team). A-team provides co-ordinated interventions that promote rational use of AMD. To date, no study has been carried out in which A-team from hospital environment goes to primary health care for the purpose of rationalization prescribing of AMD by primary health care practitioners. Project for implementation of hospital A-team in primary health care in Koprivnica-Križevci County was initiated using academic detailing method aimed at rationalization of the consumption of AMD.

ELIGIBILITY:
Inclusion Criteria:

* All primary care physicians in Koprivnica Križevci County that agree to participate in the study

Exclusion Criteria:

* Primary care physicians outside Koprivnica Križevci County

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of antimicrobials expressed as DDD per day for ATC group J01 associated with acute respiratory tract infections | 1 year
  Rationalization of consumption of antimicrobials for acute respiratory tract infections (for associated ICD diagnoses J01, J02, J03, J06, J20)

SECONDARY OUTCOMES:
Change in Clostridiodes dificile infection for patients on antimicrobial therapy | 1 year
  Number of Clostridiodes dificile infection for patients on antimicrobial therapy. A case of Clostridioides difficile infection (CDI) is defined as diarrhoeal stools or toxic megacolon and a positive laboratory assay for C. difficile toxin A and/or B in stools or a toxin-producing C. difficile organism detected in stool via culture or other means e.g. a positive PCR result.

CONTACTS AND LOCATIONS:
Overall Officials: Darija Kuruc Poje, Principal Investigator — General Hospital Koprivnica
Locations (1):
- Koprivnica križevci county, Koprivnica, Koprivnica-Križevci County, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Just IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Bryce A, Hay AD, Lane IF, Thornton HV, Wootton M, Costelloe C. Global prevalence of antibiotic resistance in paediatric urinary tract infections caused by Escherichia coli and association with routine use of antibiotics in primary care: systematic review and meta-analysis. BMJ. 2016 Mar 15;352:i939. doi: 10.1136/bmj.i939. PMID 26980184
- [Background] Costelloe C, Metcalfe C, Lovering A, Mant D, Hay AD. Effect of antibiotic prescribing in primary care on antimicrobial resistance in individual patients: systematic review and meta-analysis. BMJ. 2010 May 18;340:c2096. doi: 10.1136/bmj.c2096. PMID 20483949
- [Background] Marquet K, Liesenborgs A, Bergs J, Vleugels A, Claes N. Incidence and outcome of inappropriate in-hospital empiric antibiotics for severe infection: a systematic review and meta-analysis. Crit Care. 2015 Feb 16;19(1):63. doi: 10.1186/s13054-015-0795-y. PMID 25888181
- [Background] Teillant A, Gandra S, Barter D, Morgan DJ, Laxminarayan R. Potential burden of antibiotic resistance on surgery and cancer chemotherapy antibiotic prophylaxis in the USA: a literature review and modelling study. Lancet Infect Dis. 2015 Dec;15(12):1429-37. doi: 10.1016/S1473-3099(15)00270-4. Epub 2015 Oct 22. PMID 26482597
- [Background] Bassetti M, Righi E. Development of novel antibacterial drugs to combat multiple resistant organisms. Langenbecks Arch Surg. 2015 Feb;400(2):153-65. doi: 10.1007/s00423-015-1280-4. Epub 2015 Feb 11. PMID 25667169
- [Background] Gundlapalli AV, Beekmann SE, Graham DR, Polgreen PM; Members of the Emerging Infections Network. Antimicrobial Agent Shortages: The New Norm for Infectious Diseases Physicians. Open Forum Infect Dis. 2018 Apr 23;5(4):ofy068. doi: 10.1093/ofid/ofy068. eCollection 2018 Apr. PMID 29732380
- [Background] Nellums LB, Thompson H, Holmes A, Castro-Sanchez E, Otter JA, Norredam M, Friedland JS, Hargreaves S. Antimicrobial resistance among migrants in Europe: a systematic review and meta-analysis. Lancet Infect Dis. 2018 Jul;18(7):796-811. doi: 10.1016/S1473-3099(18)30219-6. Epub 2018 May 17. PMID 29779917
- [Background] Chitnis AS, Holzbauer SM, Belflower RM, Winston LG, Bamberg WM, Lyons C, Farley MM, Dumyati GK, Wilson LE, Beldavs ZG, Dunn JR, Gould LH, MacCannell DR, Gerding DN, McDonald LC, Lessa FC. Epidemiology of community-associated Clostridium difficile infection, 2009 through 2011. JAMA Intern Med. 2013 Jul 22;173(14):1359-67. doi: 10.1001/jamainternmed.2013.7056. PMID 23780507
- [Background] Avorn J, Soumerai SB. Improving drug-therapy decisions through educational outreach. A randomized controlled trial of academically based "detailing". N Engl J Med. 1983 Jun 16;308(24):1457-63. doi: 10.1056/NEJM198306163082406. PMID 6406886
- [Background] Soumerai SB, Avorn J. Principles of educational outreach ('academic detailing') to improve clinical decision making. JAMA. 1990 Jan 26;263(4):549-56. PMID 2104640
- [Background] O'Brien MA, Rogers S, Jamtvedt G, Oxman AD, Odgaard-Jensen J, Kristoffersen DT, Forsetlund L, Bainbridge D, Freemantle N, Davis DA, Haynes RB, Harvey EL. Educational outreach visits: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD000409. doi: 10.1002/14651858.CD000409.pub2. PMID 17943742
- [Background] Meeker D, Linder JA, Fox CR, Friedberg MW, Persell SD, Goldstein NJ, Knight TK, Hay JW, Doctor JN. Effect of Behavioral Interventions on Inappropriate Antibiotic Prescribing Among Primary Care Practices: A Randomized Clinical Trial. JAMA. 2016 Feb 9;315(6):562-70. doi: 10.1001/jama.2016.0275. PMID 26864410
- See also: WHO Antimicrobial resistance — https://www.who.int/en/news-room/fact-sheets/detail/antimicrobial-resistance
- See also: Antimicrobial Resistance: Tackling a crisis for the health and wealth of nations. The Review on Antimicrobial Resistance — https://amr-review.org/
- See also: Prioritization of pathogens to guide discovery, research and development of new antibiotics for drug-resistant bacterial infections, including tuberculosis — https://apps.who.int/iris/handle/10665/311820?locale-attribute=pt&
- See also: Antimicrobial consumption - Annual Epidemiological Report for 2017 — https://www.ecdc.europa.eu/en/publications-data/antimicrobial-consumption-annual-epidemiological-report-2017
- See also: Global Action Plan on Antimicrobial Resistance. — http://www.wpro.who.int/entity/drug_resistance/resources/global_action_plan_eng.pdf,